CLINICAL TRIAL: NCT03323177
Title: Long Term Effects of Nutritional Supplementation on Final Height of Short and Lean Adolescents: Follow-up Study to One-year Double-blind, Randomized, Placebo Controlled Studies to Evaluate the Effect of Nutritional Supplementation on Growth of Short and Lean Adolescent Boys and Girls
Brief Title: Long Term Effects of Nutritional Supplementation on Final Height
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: finally it was decided not to initiate the study due to logistical issues
Sponsor: Rabin Medical Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RMC025117ctil
Record Dates: First submitted 2017-10-03; First posted 2017-10-26 (Actual); Last update posted 2019-12-27 (Actual); Status verified 2018-04

CONDITIONS: Growth Disorders; Low Weight; Short Stature
MeSH Terms: conditions — Growth Disorders; Thinness; Dwarfism

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nutritional supplementation gender specific formula (Experimental): Patients at this arm will continue to consume the study formula until final height. The formula is a gender specific powder added to water containing about 25% of recommended Daily Recommended Intake (DRI) for calories, high protein (25% of calories) and multi vitamin and mineral (255-100%) of DRI for recommended daily allowance (RDA) or adequate intake
  Interventions: Dietary Supplement: Gender specific nutritional standardized formula
- Follow-up only (Other): Patients who are reluctant to continue to consume the study formula will come to follow-up visits only without any intervention until final height is reached
  Interventions: Other: Follow-up only

INTERVENTIONS:
Dietary Supplement: Gender specific nutritional standardized formula — Patients will continue to consume the study formula until final height: gender specific powder added to water containing about 25% of recommended DRI for calories, high protein (25% of calories) and multi vitamin and mineral (255-100%) of DRI for recommended daily allowance (RDA) or adequate intake
  Arms: Nutritional supplementation gender specific formula
Other: Follow-up only — Patients who are reluctant to continue to consume the study formula will come to follow-up visits only without any intervention until final height is reached
  Arms: Follow-up only

SUMMARY:
The proposed study is an extension study to two ongoing double blind, randomized, placebo-controlled studies evaluating the effect of gender-specific nutritional supplementation on growth of short and lean adolescent boys and girls. The aim of the current study is to extend these short term double blind, randomized, placebo controlled studies (one in boys and one in girls) and to add an extension study, which will evaluate the long term effect of the gender specific nutritional supplementation on final height. Patients completing the ongoing studies will be offered to continue treatment with the study formula until final height. Patients reluctant to continue to consume the study formula will be offered to continue followup only during the extension study without any intervention.

ELIGIBILITY:
Inclusion Criteria:

* Participation in the former double blind, randomized, placebo controlled study to evaluate the effect of nutritional supplementation on growth of short and lean adolescent boys (protocol no. 0676-14) and girls (protocol no. 0002-15).
* Completing at least the double blind phase of the previous studies (protocol no 0676- 14 or 0002-15)
* Signing informed consent forme

Exclusion Criteria:

* Diagnosis of Growth Hormone Deficiency or treatment with Growth Hormone
* Any known chronic disease or dysmorphic syndrome including: bone diseases, organic brain diseases, neurological disease, past or current malignancy, chronic cardiac, renal or pulmonary problems
* Any known gastrointestinal disease including malabsorption
* Any known organic reason for growth retardation
* Any chronic treatment with medication that might affect appetite, weight or growth

Ages: 10 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2018-06 (Estimated); Primary Completion 2022-06 (Estimated); Study Completion 2022-06 (Estimated)

PRIMARY OUTCOMES:
Final Height Standardized Deviation Score (SDS) | Up to 7 years (after reaching final height:height velocity less than 1 centimeter per year)

SECONDARY OUTCOMES:
Weight Standard Deviation Score | Up to 7 years (after reaching final height:height velocity less than 1 centimeter per year)
Body Mass Index (BMI) Standard Deviation Score | Up to 7 years (After reaching final height: height velocity less than 1 centimeter per year)
Duration of puberty | Up to 7 years (After reaching full puberty:tanner stage 5)
  Duration of Puberty (in Years ) from tanner stage 2 until reaching tanner stage 5
Quality of Life | Up to 7 years (After reaching final height:height velocity less than 1 centimeter per year)
  Quality of life as measured through Quality of Life Questionnaire
Self Esteem | Up to 7 years (After reaching final height:height velocity less than 1 centimeter per year)
  Self Esteem as measured through Self Esteem Questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Schneider Children's Medical Center, Petah Tikva, Israel